CLINICAL TRIAL: NCT04027959
Title: Novel Skin Preparation Approaches for Transdermal Delivery by Iontophoresis of a Low Molecular Weight, Positively Charged Compound (Vitamin B12) to the Systemic Circulation
Brief Title: Transdermal Iontophoresis of Vitamin B12 Under Three Different Skin Preparations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mark A. Kortsen, MD, Gastroenterology Senior Consultant, James J. Peters Veterans Affairs Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: KOR-17-34
Record Dates: First submitted 2019-07-19; First posted 2019-07-22 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Macrocytic Anemia With Vitamin B12 Deficiency
Keywords: Transdermal Penetration Enhancers, Iontophoresis, Neostigmine, Glycopyrrolate, Vitamin B12, Methylcobalamin, Cyanocobalamin
MeSH Terms: interventions — Vitamin B 12; Iontophoresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Epilation (Experimental): Hair epilated prior to application of Vitamin B12 solution to skin
  Interventions: Dietary Supplement: Vitamin B12
- Oleic Acid (Experimental): Oil is allowed to soak the skin prior to application of Vitamin B12 solution to skin
  Interventions: Dietary Supplement: Vitamin B12
- No Prep (Experimental): Skin is cleansed with an alcohol wipe prior to application of Vitamin B12 solution to skin
  Interventions: Dietary Supplement: Vitamin B12

INTERVENTIONS:
Dietary Supplement: Vitamin B12 — Diffusion of Vitamin B12 through the skin over 20 minutes under the effect of low amount of direct electric current
  Other Names: Iontophoresis

SUMMARY:
STUDY DESIGN: Phase I Clinical Trial The researchers set out to assess the effectiveness of transdermal iontophoretic administration of Vitamin B12 (V.B12) under three different skin preparatory conditions.

SETTING: James J. Peters Veterans Affairs Medical Center (Bronx, NY) BACKGROUND: Poor skin permeability precludes the use of transdermal route from being used in common clinical practice for rapid and precise administration of medications through intact skin that are expected to have a systemic effect. The researchers determined the relative effectiveness of an unconventional transdermal iontophoresis technique for the administration of Vitamin B12 (V.B12) under three different skin preparatory conditions.

METHODS: During this study, Vitamin B12 (V.B12) was administered through the skin of volunteer human research subjects. Iontophoresis was used as transdermal medication delivery modality after pre-treatment of the skin in 3 different ways. The sequence of skin preparations was arranged in a random order for each subject. Method 1 was called "No Prep", serving as the control approach; method 2 was called "Oleic Acid" application to the skin for 40 minutes; and method 3 was hair "Epilation" (e.g. hair removal by plucking). Fifteen milligrams of aqueous solution of V.B12 was administered through intact, previously unused skin of an anterior thigh during all 3 tests. Chemoluminescence, on an automated laboratory reader Advia Centaur-XP, was used to determine the serum concentration of V.B12 prior to and after transdermal iontophoretic delivery. All 3 experiments were performed on the same day within an hour of each other. The subject's blood was drawn prior and 10 minutes after the 20-minute long sessions of transdermal V.B12 iontophoresis. We were able to calculate the increase in serum V.B12 concentration and based on estimated blood volume, the total quantity and percent dose delivered systemically.

DETAILED DESCRIPTION:
In order to quantify the changes in skin permeability to drugs delivered by ION under three different preparatory conditions, we used V.B12 as a model substance. Its choice was dictated by its inherent safety, positive charge and quantification of serum concentration readily available through our clinical laboratory. We compared the effects of unprepared skin (No Prep), oil-soaked skin [ref. 9-12] (Oleic Acid) and skin from which hair have been plucked out of (Epilation), on the serum concentrations of V.B12 before and after administration via ION.

Veterans and non-Veterans without SCI were recruited for the study comparing the three skin preparation methods. This prospective, skin preparatory method sequence-randomized study was approved by the Institutional Review Board of the James J. Peters VA Medical Center (JJPVAMC). The ION equipment used was a standard FDA-approved wired ION controller unit (IBOX by Dynatronics) and 4mL ION electrodes by (ionto+ by Richmar). The skin was prepared using 1 of the 3 techniques, performed in a random order. Each subject was assigned a 2-digit sequential number. A random-numbers table was used to assign the sequence of methods to each subject. A single positive electrode patch containing 4mL of a water-based solution with 15mg of V.B12 was used per experiment. One negative electrode patch was also used to complete the circuit. Blood was drawn prior to the first administration. Thirty minutes after the start of the ION delivery of the V.B12 through the skin of anterior thigh, the blood was drawn again. The blood was centrifuged for 5 minutes and delivered to the clinical laboratory for testing without delay. Serum concentration of V.B12 was measured using chemoluminescence on an automated laboratory reader Advia Centaur-XP. The experiments were conducted sequentially in a timely fashion, performed on the same day and within a span of 3 hours. Blood was drawn for a total of 4 times per subject.

The "No Prep" technique was performed by simply wiping the two skin surfaces on an anterior thigh, where the electrodes were later attached, with two-70% isopropyl alcohol prep. pads. The skin surface destined for positive electrode application was sprayed with a thin layer of 20% Benzocaine (Americaine aerosol spray can) and covered with an occlusive plastic film for 10 minutes. The film was then removed and the skin was cleansed with water-moistened paper towel, followed by one alcohol prep. pad.

The "Oleic Acid" technique involved first wiping the two skin patches and later soaking the skin patch, where the positive electrode was going to be placed, with oil called oleic acid for 40 minutes. The oil was then wiped off with a paper napkin and an alcohol pad. That same skin area was sprayed with a thin layer of 20% Benzocaine (Americaine aerosol spray container) and covered with an occlusive plastic film for 10 minutes. The film was then removed and the skin was cleansed with water-moistened paper towel, followed by one alcohol prep.

The "Hair Epilation" technique involved first wiping the two skin patches with 2-70% isopropyl alcohol skin preps and sprayed with a thin layer of 20% Benzocaine (Americaine aerosol spray container) and covered with an occlusive plastic film for 10 minutes. The film was removed and the skin was cleansed with de-ionized water followed by alcohol prep. Hair removal, using an epilator machine (Remington EP 7030), was performed by clearing an area of 5x5cm or 2x2 inch square. The epilated area was then covered with a thin layer of 0.2% Sodium Lauryl Sulfate (SLS) in de-ionized water.

After each of the skin preparations and without delay, 15mg of methylcobalamin dissolved in 4mL of de-ionized water soaked into the anode patch reservoir was applied to the designated skin of the proximal anterior thighs. The 7x7cm skin area under the negative electrode was wiped with an alcohol pad and 0.5mL of 1% citric acid dissolved in 0.9% normal saline solution was applied to the negative electrode's skin contact surface. The return (negative) electrode was then attached to the skin 10cm from the positive electrode.

An elevated room temperature of 73-78 degrees Fahrenheit (25 degrees Celsius) was maintained in the room for the purposes of maintaining adequate blood flow in the peripheral dermal capillaries. No exclusion criteria for diseases that decrease capillary perfusion such as diabetes have been utilized. As a result, 2 of the 10 subjects who participated in this study had a diagnosis of Diabetes Mellitus type 2.

IBOX ION device was attached to the electrodes by way of wire leads and a multimeter was attached to the electrodes in parallel in order to record the skin's electrical resistivity prior to and after ION. Throughout the 20-minute ION session, voltage exerted by the IBOX was recorded at regular intervals. The voltage was automatically adjusted by the IBOX to deliver a pre-set constant electrical current of 4mA/minute. Throughout the procedure subjects were asked about the presence of any sensations associated with the ION including effects of the medication being administered.

ELIGIBILITY:
Inclusion Criteria:

* Able-bodied,
* Male or female,
* Between the ages of 18-80 years old.

Exclusion Criteria:

* Previous adverse reaction or hypersensitivity to electrical stimulation,
* Pregnancy (women who are sexually active and of childbearing potential must utilize a method of contraception and agree to maintain a contraceptive method until completion of the study),
* Inability to provide informed consent,
* History of ingrown hair folliculitis after shaving or epilation,
* Allergy to Sodium Lauryl Sulfate, Oleic acid, Silver Chloride, Agarose Gel, Methylcobalamin, Citric Acid, Isopropyl alcohol, Benzocaine, Polyethylene film, Polyethylene Glycol solvent,
* Concurrent illness with fever,
* Concurrent participation in a research study,
* VA employee.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Amount of Vitamin B12 delivered into the systemic circulation | 20 minutes
  micrograms

CONTACTS AND LOCATIONS:
Overall Officials: Mark Korsten, MD, Principal Investigator — Employee
Locations (1):
- James J Peters VA Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD information